CLINICAL TRIAL: NCT03307850
Title: Feasibility Study to Assess the Impact of Non-glucose Signals on Glycemic Control in Patients With Type 1 Diabetes on Sensor Augmented Insulin Pump
Brief Title: Impact of Non-glucose Signals on Glycemic Control in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Mayo Clinic (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JDRFSignals1
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes; hypoglycemia; exercise; stress; artificial pancreas; cortisol
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation of Exercise (Experimental): Observation During Exercise and Stress
  Interventions: Other: Observation During Exercise and Stress

INTERVENTIONS:
Other: Observation During Exercise and Stress — Patients with type 1 diabetes (T1D) on an insulin pump will be studied for 5 weeks in the outpatient setting performing their normal activities, to include their normal diet and exercise, while assessing the amount of type of exercise performed, and emotional stress levels, using stress sensor, questionnaires and salivary cortisol levels.
  Subjects at the William Sansum Diabetes Center will perform graded exercise on a treadmill for up to 45 minutes with all activity and stress monitors running, achieving 30 and 60% calculated heart rate reserve, once during the study. Subjects at Mayo Clinic will perform a graded exercise test on a treadmill to determine V02max and ensure stable cardiac status, once during the study.

SUMMARY:
This clinical trial will identify exercise-related and emotional stress related effects on glycemic control in patients with type 1 diabetes using sensor-augmented pump (SAP) therapy.

DETAILED DESCRIPTION:
Patients with type 1 diabetes (T1D) on an insulin pump will be studied for 5 weeks in the outpatient setting performing their normal activities, to include their normal diet and exercise, while assessing the amount of type of exercise performed, and emotional stress levels, using stress sensor, questionnaires and salivary cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Clinical diagnosis, based on investigator assessment, of T1D for at least one year and using insulin for at least 1 year.
* Using an insulin pump for diabetes therapy for at least 3 months
* Demonstration of proper mental status and cognition for the study
* Non-smoker
* If not currently using CGM, willing to use CGM during the study
* An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

* Admission for diabetic ketoacidosis in the 6 months prior to enrollment unless study team feels the subject is appropriate for study given complete clinical context for subject
* Severe hypoglycemia resulting in seizure or loss of consciousness > once in the 6 months prior to enrollment
* History of a seizure disorder (except hypoglycemic seizure), unless written clearance is received from a neurologist and not currently on a seizure medication
* Cystic fibrosis
* Unstable coronary artery disease or heart failure, unless written clearance is received from a cardiologist or primary care provider
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  1. Inpatient psychiatric treatment in the past 6 months
  2. Presence of a known adrenal disorder or chronic oral steroid therapy
  3. Abnormal liver function test results (Transaminase >3 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
  4. Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2);
  5. Active gastroparesis (defined actively being treated with medications)
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
* Abuse of alcohol or recreational drugs
* Pregnancy
* Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis).
* Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg) at the time of screening
* Uncontrolled microvascular complications such as current active proliferative diabetic retinopathy defined as proliferative retinopathy requiring treatment (e.g. laser therapy) in the past 12 months.
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Impact of Stress and Exercise on CGM Glucose Levels, determining how these factors affect time within target glucose range 70-180 mg/dl | 5 Weeks
  Examine the impact of Stress and Exercise on CGM Glucose Levels, determining how these factors affect time within target glucose range 70-180 mg/dl. Correlate these factors that influence glycemic control to inform future algorithm development for an artificial pancreas (AP) device to better handle exercise and stress related events to be used in a future study.

SECONDARY OUTCOMES:
CGM Glucose Levels 70-180 mg/dl | 5 Weeks
  CGM Glucose Levels, within target range 70-180 mg/dl
CGM Glucose Levels less than 70 mg/dl | 5 Weeks
  CGM Glucose Levels, less than 70 mg/dl
CGM Glucose Levels greater than 180 mg/dl | 5 Weeks
  CGM Glucose Levels, greater than 180 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Yogish C Kudva, MD, Principal Investigator — Mayo Clinic; Eyal Dassau, PhD, Principal Investigator — Harvard University; Jordan E Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (2):
- United States (2):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No